CLINICAL TRIAL: NCT07242859
Title: Effects of Rice Bran on Radiation-Induced Oral Mucositis in Patients With Head/Neck Cancer and Its Impact on the Quality of Life
Brief Title: Rice Bran Supplementation for Radiation-Induced Oral Mucositis in Head and Neck Cancer
Acronym: RICE-MUC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Milad Lobos (Other)
Responsible Party: Sponsor-Investigator, Christina Milad Lobos, Sponsor-Investigator, Assistant Lecturer, German University in Cairo
Organization: German University in Cairo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-2025-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Radiation-Induced Oral Mucositis; Head &Amp; Neck Cancer; Head &Amp; Neck Squamous Cell Carcinoma
Keywords: Radiation-Induced Oral Mucositis; Oral Mucositis; Head and Neck Cancer; Rice Bran; Dietary Supplement; Radiation Therapy Side Effects; Quality of Life; Supportive Care; Antioxidants; Cancer Treatment Support
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: This is a parallel-group interventional study where participants are assigned to one of two groups. The active group receives rice bran supplements during radiation therapy, while the control group receives standard care without rice bran. The study compares the effects of rice bran on radiation-induced oral mucositis and quality of life between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rice Bran Supplement Group (Experimental): Participants in this group will receive rice bran supplements daily during their radiation therapy. The supplement is intended to reduce the severity of oral mucositis and improve quality of life.
  Interventions: Dietary Supplement: rice bran
- Control Group (Standard Care) (No Intervention): Participants in this group will receive standard care during radiation therapy without rice bran supplementation. Their oral mucositis symptoms and quality of life will be monitored for comparison.

INTERVENTIONS:
Dietary Supplement: rice bran — Participants in the intervention group will receive a standardized dose of rice bran supplement administered orally each day throughout the course of their radiation therapy. The rice bran used is a natural dietary supplement rich in antioxidants and anti-inflammatory compounds, aimed at reducing the severity and duration of radiation-induced oral mucositis in patients with head and neck cancer.
  Other Names: Oryza
  Arms: Rice Bran Supplement Group

SUMMARY:
This study aims to find out if taking rice bran supplements can help reduce the painful mouth sores (oral mucositis) that often occur in patients with head and neck cancer who receive radiation therapy. The trial will include adult patients undergoing radiation treatment. Participants will be given rice bran supplements during their therapy to see if it can lessen these side effects and improve their overall quality of life.

DETAILED DESCRIPTION:
Radiation-induced oral mucositis is a common and debilitating side effect experienced by patients undergoing radiation therapy for head and neck cancer. This condition causes painful inflammation and ulceration of the mucous membranes in the mouth, significantly impacting patients' ability to eat, speak, and maintain oral hygiene, thereby reducing their quality of life.

This study investigates the therapeutic potential of rice bran, a natural byproduct of rice milling rich in antioxidants and anti-inflammatory compounds, as a dietary supplement to mitigate the severity of oral mucositis. Participants will be adult patients diagnosed with head and neck cancer who are scheduled to receive radiation therapy.

The intervention involves administering rice bran supplements concurrently with radiation treatment. The study aims to evaluate the effects of rice bran on the incidence, duration, and severity of oral mucositis, as well as its overall impact on patients' quality of life during and after treatment.

By assessing clinical outcomes and patient-reported measures, this trial seeks to provide evidence on whether rice bran can serve as an effective, low-cost, and accessible supportive care option for managing radiation-induced oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of age 18 years old tor more
* Patients with squamous cell carcinomas without metastases of other non-head and non-neck tumors.
* Patients undergoing radiotherapy with an ECOG performance status of 0, 1, or 2
* Patients who will receive IMRT delivered as radical or adjuvant therapy with or without concurrent chemotherapy
* Ready to provide written informed consent

Exclusion Criteria:

* Receiving any other approved or investigational anti-cancer agent than those specified in this study.
* Pregnant or breastfeeding female patients
* Patients who have oral lesions unrelated to treatment or cancer,
* Patients who are on drugs that could cause oral lesions or are using anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 mucositis . | From the start of radiation therapy until 2 weeks after completion of treatment (approximately 8 weeks)
  The proportion of patients who develop severe oral mucositis of grade 3 or higher, based on standardized clinical grading scales, during or after radiation therapy. Grade 3 mucositis is characterized by severe pain, ulceration, and an inability to eat solid foods without significant discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- German university in cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No